CLINICAL TRIAL: NCT03961620
Title: Prospective Observational Study on the Incidence of Perioperative Hypothermia and the Effect of Standard Normothermia Measures at the Surgical Area of Parc Tauli Hospital Universitari, Sabadell: Tauli-Previnq-Warm
Brief Title: Study on the Incidence of Perioperative Hypothermia at the Surgical Area of Parc Tauli Hospital Universitari, Sabadell
Acronym: PREVINQ-WARM
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: 3M (Industry)
Responsible Party: Principal Investigator, Xavier Guirao, Coordinator of Endocrine, Head and Neck Surgery Unit, Corporacion Parc Tauli
Other Study IDs: 2018/630
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Hypothermia
Keywords: perioperative hypothermia; core temperature; perioperative normothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: The SpotOn system that encompasses the registration unit (3M SpotOn Control Unit), disposable sensor (3M SpotOn Control Sensor) along with the cords and electric power unit. — Patients submitted to major surgical procedure will be assessed for core body temperature by employing SpotOn sensor device, before, during and after surgical procedure.

SUMMARY:
The study TAULÍ-PREVINQ-WARM will assess the rate of perioperative hypothermia in patients submitted to major surgical procedures at the operating room main area (and at the ambulatory surgery building for ophthalmologic major procedures) of the Parc Taulí, Hospital Universitari, Sabadell, Barcelona.

DETAILED DESCRIPTION:
Treatment plan The month before the start of the study, investigators will double check with the administrative personnel the potential candidates to be included in to the study. Furthermore, investigators will meet with the responsible of each surgical specialty to delineate the adequate staff workload and collaborators needs. To assure the best study performance and to avoid selection patient bias, patients will be consecutively included in blocs of each designated surgical specialty.

At the patient admission area and surgical preparation, associated investigators will inform to candidates and relatives about the project giving the informed form to be signed.

Patient inclusion will include a pilot phase (four to five patients) to teach collaborators regarding the correct placement of cutaneous sensor, data lecture and registration to the database. Along with the maintenance department of the hospital, we also assess the correct installation and function of temperature and humidity sensors at the OR (Mini-datalogger 174H, Instrumentos Testo, S.A. Cabrils, Barcelona). OR temperature and the degree of humidity will be measured at the specific time points stated at the paragraph of the measurements.

Body temperature (BT) measurements will be performed at the UPQ, anesthesia preparation room, OR and URPA in those specifically stated time points (Annex 2 and Figure 1).

Because the investigators want to perform a pragmatic study, patients will receive conventional normothermia preventive measures following the approved local guidelines from the Anesthesiology Department.

Measurement and data entry Body temperature (BT) Patient's BT will be assessed with the SpotOn system that encompasses the registration unit (3M SpotOn Control Unit), disposable sensor (3M SpotOn Control Sensor) along with the cords and electric power unit.

Non-invasive digital BT system monitorization SpotOn, includes a sensor that by adhering to the lateral side of supra-ocular region, allows for continued registration of BT for the overall surgical process.

Number of times and sites of BT registration Staff devoted to assess BT measurements. Staff from 3M, will advise nurses, anesthesiologists and investigators regarding SpotOn specifications and management at the beginning of the study

Because OR temperature and degree of humidity may have some influence on patient's BT and thermic comfort both patients and OR staff, OR temperature and humidity will be registered at the beginning and at the end of surgical procedure. Also, the protocol will take in to the account weather conditions registered at the MeteoCat and will be included at the data base regularly. Also, staff from Maintenance of Hospital Facilities and Equipment, will set up and store data from the OR temperature and humidity sensors (Mini-datalogger 174H, Instrumentos Testo, S.A. Cabrils, Barcelona).

Data about measures addressed to sustain perioperative normothermia will also be recorded (see Annex 4)

At the end of surgical procedure the investigators will ask patients and OR staff for running a visual analogic scale punctuation (1 to 10) regarding the perceived thermal comfort (see Annex 5)

Length of the study and period of patients recruitment. Because the specific nature of this prospective observational and pragmatic study, the rate of patients recruitment will be assessed frequently to accommodate both optimal patient accrual and fair and adequate entry data. The approximate time for total patients inclusion will be of one year.

Sample size The main objective of the study TAULI-PREVINQ-WARM is to assess the rate of perioperative hypothermia (<36ªC) at some point during the surgical process in patients operated on for a major surgical procedure at the Parc Tauli, Hospital Universitari, Sabadell. Then, sample size has been calculated taking in to the account that roughly 50% of patients will have some kind of hypothermia with 10% of variability of 95% CI. Assuming a10% of repository additional patients, 110 patients will be included overall.

Assessment of data results and statistical analysis. The TAULI-PREVINQ-WARM is a pragmatic study that wants to assess body temperature in surgical patients under regular clinical conditions. We will perform a descriptive analysis of data by depicting mainly frequency distribution analysis of the qualitative main variable, HypoTer. The proposed sample size will allow also for assessing the rate HypoTer at each different surgical areas where patients are admitted. Also, repeated measures will be compared among different surgical procedures at the OR taking in to consideration the body surface area under regular preventive normothermia measures, following the general lineal model. Univariate two-sided analysis will be perform for all comparisons and parametric or non-parametric analysis will be performed accordingly. Multivariate analysis might eventually be performed depending of the rate of events.

ELIGIBILITY:
Inclusion Criteria:

* ASA score I to IV
* Patients submitted to major surgical procedures at the main OR facilities (or at the ambulatory surgery building for ophthalmologic procedures) under general or neuraxial anesthesia from surgical specialties
* Patients (parents or legal guardians regarding pediatric patients) that have signed informed consent form.

Exclusion Criteria:

* Patients submitted to craniofacial neurosurgical procedures
* Patients submitted to any surgical procedure requiring draping or sterile isolation of the frontal part of head, precluding intraoperative assessment of SpotOn sensor.
* Patients (parents or legal guardians regarding pediatric patients) that have not signed informed consent form.
* Patients that by the time of the hospital admission present a relevant inflammatory or infectious process at the skin of frontal part of the head
* Patients diagnosed with psychiatric disease relevant enough to avoid adequate staff-patients communication for this specific study

Ages: 8 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients submitted to elective major surgical procedures from different surgical specialties
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Rate of perioperative hypothermia (<36ºC) | 12 hours
  Body temperature measured by SpotOn system sensor in different surgical procedures and at any specific surgical area.

SECONDARY OUTCOMES:
Type and duration of applied physical measures to prevent periopertive hypothermia | 12 hours
  The investigators will corroborate whether or not textile blankets, forced air warming blankets or additional measures are applied, anf if so, the time and durations of such measures.
Temperature at the operating room | 1-6 hours
  Temperature and degree of humidity at the OR
Thermal confort | 1-6 hours
  Thermal comfort of patients and OR staff members
Adverse events | Up to 30 days (1 year for prosthetic surgery)
  Rate of postoperative adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Guirao, MD, Principal Investigator — Parc Tauli Hospital Universitari, Sabadell
Locations (1):
- Parc Tauli Hospital Universitari, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No